CLINICAL TRIAL: NCT02638909
Title: A Phase II, Multicenter, Single-Arm Study of Oral Ceritinib in Adult Patients With ALK and ROS1 Activated Gastrointestinal Malignancies
Brief Title: Study of Oral Ceritinib in Patients With ALK and ROS1 Activated Gastrointestinal Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Criterium, Inc. (Industry)
Collaborators: University of Colorado, Denver (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOV-ALK-01
Record Dates: First submitted 2015-12-15; First posted 2015-12-23 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Adenocarcinoma; Cholangiocarcinoma; Pancreatic Adenocarcinoma; Hepatocellular Adenocarcinoma; Gastric Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: Gastrointestinal malignancies
MeSH Terms: conditions — Cholangiocarcinoma; Adenocarcinoma Of Esophagus | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ceritinib (Experimental): Phase II, single-arm study of oral ceritinib in adult patients with ALK and ROS1 activated gastrointestinal malignancies
  Interventions: Drug: ceritinib

INTERVENTIONS:
Drug: ceritinib — Treatment with ceritinib will continue until patient experiences unacceptable toxicity that precludes further treatment, discontinues treatment at the discretion of the investigator or patient, starts a new anticancer therapy and/or dies.
  Other Names: Zykadia

SUMMARY:
The available data indicate that Ceritinib has substantial anti-tumor activity in patients with anaplastic lymphoma kinase (ALK) and ROS1 rearranged non-small cell lung cancer (NSCLC). This trial will investigate the potential of Ceritinib in patients with advanced gastrointestinal malignancies with ALK and ROA1 rearrangement, and for whom there is no available therapeutic option.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter, phase II study of ceritinib in adult patients with ALK- and ROS1 activated colorectal, cholangiocarcinoma, pancreatic, hepatic, gastric, or esophageal adenocarcinoma. An estimated 500 patients will be screened for ALK and ROS1 by fluorescence in situ hybridization (FISH) and immunohistochemistry (IHC) per institutional standard of care (SOC), and/or ALK/ROS1 by next-generation sequencing (NGS). At least 30 identified patients will be treated with ceritinib per protocol. Treatment with ceritinib will continue until patient experiences unacceptable toxicity that precludes further treatment, discontinues treatment at the discretion of the investigator or patient, starts a new anticancer therapy and/or dies.

Male and female patients aged 18 or over that have colorectal adenocarcinoma, cholangiocarcinoma, pancreatic, hepatocellular, gastric or esophageal adenocarcinoma that contain an activated ALK gene due to rearrangement, mutation, amplification, translocation or other mechanisms. Patients must have been pretreated with cytotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of inoperable colorectal adenocarcinoma, pancreatic, hepatocellular, cholangiocarcinoma, small bowel, gastric or esophageal adenocarcinoma that carries an activated ALK or ROS1 pathway
2. Age 18 years or older at the time of informed consent.
3. Patients must have received at least 1 line of cytotoxic chemotherapy
4. Patients must have archival tissue sample available, collected either at the time of diagnosis or any time since.

   - If archival tissue is unavailable, patient must be eligible and willing to undergo a fresh tissue biopsy
5. Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 2 (CTCAE v 4.03) provided that concomitant medication is given prior to initiation of treatment with LDK378, except for patients with grade 2 nausea/vomiting and/or grade 2 diarrhea despite optimal supportive therapy who will not be allowed to participate in the study. Additionally, patients with any grade of alopecia are allowed on treatment.
6. Cohort Expansion Phase: Patient must have measurable lesions as defined by RECIST version 1.1 criteria.
7. ECOG performance status 0-2
8. Patients must have normal organ and marrow function as defined below: Bone marrow function defined as the following: An absolute neutrophil count ≥ (ANC) 1,500/mcl. Platelets ≥ 75,000/mcl. Hemoglobin ≥ 8 g/dl.
9. Renal function defined as the following: Serum creatinine less than or equal to 1.5 x institutional upper limit normal (ULN). Calculated or measured creatinine clearance (CrCL) ≥ 30 mL/min
10. Hepatic function defined as the following: Serum total bilirubin < 1.5 x ULN. AST (SGOT), ALT (SGPT), and alkaline phosphatase ≤ 3.0 x ULN. Serum albumin ≥ 2.5 g/dl. If liver involvement, AST, ALT, and alkaline phosphatase ≤ 5.0 x ULN.
11. Serum amylase ≤ 2 x ULN and serum lipase ≤ 1 x ULN
12. Fasting plasma glucose ≤175 mg/dL (≤9.8 mmol/L)
13. Patient must have the following laboratory values or have the following laboratory values corrected with supplements to be within normal limits at screening:

    * Potassium ≥ lower limit of normal (LLN)
    * Magnesium ≥ LLN
    * Phosphorus ≥ LLN
    * Total calcium (corrected for serum albumin) ≥ LLN
14. A male subject of fathering potential must use an adequate method of contraception to avoid conception throughout the study [and for up to 12 weeks after the last dose of study drug] to minimize the risk of pregnancy. If the partner is pregnant or breastfeeding, the subject must use a condom. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
15. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of study drug to minimize the risk of pregnancy. WOCBP must have a negative serum or urine pregnancy test within 72 hours before the start of the investigational product. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening) with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate. For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
    * Combination of any two of the following (a+b or a+c or b+c):
    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS).

    Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.

    In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
16. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 3 weeks (4 weeks for radiotherapy to the lung fields and 6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients with known hypersensitivity to any of the excipients of ceritinib (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate)
3. Prior therapy with ceritinib or other ALK or ROS1 inhibitor agents
4. Patients who are currently receiving treatment with warfarin sodium (Coumadin®) or any other coumarin-derivative anti-coagulants.
5. Patients with symptomatic CNS metastases who are neurologically unstable or have required increasing doses of steroids within the 1 week prior to study entry to manage CNS symptoms.
6. Impairment of GI function or GI disease that may significantly alter the absorption of ceritinib
7. History of pancreatitis or history of increased amylase or lipase that was due to pancreatic disease.
8. Patients with known history of extensive disseminated bilateral interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and clinically significant radiation pneumonitis (i.e. affecting activities of daily living or requiring therapeutic intervention).
9. Cardiac conditions as follows:

   * Active coronary artery disease, unstable or newly diagnosed angina or myocardial infarction less than 6 months prior to first study drug administration.
   * Class II-IV New York Heart Association (NYHA) congestive heart failure.
   * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin
   * QTc (Frederica) prolongation > 470 msec.
   * Subjects with valvular heart disease CTCAE (Version 4.0) Grade 2.
   * Known left ventricular ejection fraction (LVEF) < 50%.
   * Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without anti-hypertensive medication
10. Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with LDK378 and for the duration of participation:

    * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (please refer to http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm)
    * Strong inhibitors or strong inducers of CYP3A4/5 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
    * Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, and/or CYP2C9 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
    * Therapeutic doses of warfarin sodium (Coumadin) or any other coumarin-derived anti-coagulant. Anti-coagulants not derived from warfarin are allowed (e.g., dabigatran, rivaroxaban, apixaban).
    * Unstable or increasing doses of corticosteroids
    * Enzyme-inducing anti-convulsive agents
    * Herbal supplements
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris (Canadian Cardiovascular Society grade II-IV despite medical therapy), cardiac arrhythmia, active bleeding diatheses, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Major surgical procedure, open biopsy, or significant traumatic injury less than 4 weeks or those who receive minor surgical procedures (e.g. core biopsy or fine needle aspiration) within 1 week from first dose of first study drug administration.
13. Known inability to swallow up to five LDK378 capsules daily.
14. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-12; Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) of ceritinib, as defined as the percentage of patients who have achieved complete response, partial response, and stable disease at 2 months per RECIST 1.1) to ceritinib by investigator assessment | 2 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 20 months
Objective tumor response based on computed tomography scans (or magnetic resonance imaging if patients are allergic to iodinated contrast) per RECIST 1.1 criteria | 2 months
  Antitumor activity of ceritinib will be based on the best overall response. Response rate (complete response [CR], partial response [PR], CR + PR) will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lieu, MD, Principal Investigator — Criterium Inc., d.b.a. Academic GI Cancer Consortium (AGICC)
Locations (6):
- United States (6):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Laura & Isaac Permutter Cancer Center at NYU Langone, New York, New York
  - The Ohio State University, James Cancer Hospital, Columbus, Ohio
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided